CLINICAL TRIAL: NCT01684761
Title: A Phase 2 Double-Blind, Placebo Controlled Multi-Center Study to Evaluate the Efficacy and Safety of Tcelna in Subjects With Secondary Progressive Multiple Sclerosis
Brief Title: Study of Tcelna (Imilecleucel-T) in Secondary Progressive Multiple Sclerosis
Acronym: Abili-T
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Opexa Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Protocol Number 2012-00
Record Dates: First submitted 2012-09-11; First posted 2012-09-13 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Autoimmune Diseases of the Nervous System; Multiple Sclerosis; Secondary Progressive Multiple Sclerosis; Disease Progression; Brain Atrophy
Keywords: Multicenter Study; Randomized Controlled Trial; Individualized Medicine; Immunotherapy; Myelin Proteins; Biological Agents
MeSH Terms: conditions — Autoimmune Diseases of the Nervous System; Multiple Sclerosis; Multiple Sclerosis, Chronic Progressive; Disease Progression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tcelna (Experimental): 30-45 x 10E6 total cells in 2 ml. Subjects receive two annual courses of 5 subcutaneous doses each year (at 0, 4, 8, 12 and 24 weeks).
  Interventions: Biological: Tcelna
- Placebo (Placebo Comparator): Tcelna inactive ingredients (without cells) totaling 2 ml per dose. Administered subcutaneously with same two year treatment regimen as experimental treatment arm.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Tcelna — Autologous pool of myelin reactive T-cells (MRTC) expanded ex vivo with immunodominant epitopes selected from the three myelin antigens, MBP, PLP and MOG on a per subject basis. Attenuated by irradiation to prevent further proliferation before releasing product for administration.
  Arms: Tcelna
Biological: Placebo — 2 ml of Tcelna excipients, prepared daily as individual doses and irradiated before releasing product for administration.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether Tcelna (imilecleucel-T, autologous T-Cell Immunotherapy) is effective in the treatment of secondary progressive multiple sclerosis (SPMS).

DETAILED DESCRIPTION:
Subjects whose myelin reactive T-cell can be identified by EPA will are randomized and provide blood to manufacture Tcelna. Approximately 5 weeks after receipt of the subject's whole blood procurement, the subjects will receive either Tcelna or placebo and will complete baseline assessments and will receive study treatments at Weeks 0, 4, 8, 12, and 24 (Visits 3-7), totaling 5 doses in year one.

Approximately one month prior to the Week 52 visit a second blood procurement will be performed and the subject will receive the second series of treatments as received in the first year study schedule. Subjects will be evaluated for changes in disability and cognitive function every 3 months, and radiographic changes annually.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with MS as defined by the modified McDonald criteria
* SPMS defined as relapsing-remitting disease with recent progression in MS-related neurological deficits
* EDSS score 3.0 - 6.0, inclusively
* Presence of myelin reactive T-cells

Exclusion Criteria:

* Diagnosed with primary progressive MS
* Treatment with beta-interferon, glatiramer acetate or dimethyl fumarate 30 days prior to screening
* Treatment with ACTH, any over-the-counter or prescription corticosteroids 60 days prior to screening
* Treatment with IVIG, plasmapheresis or cytopheresis 90 days prior to screening
* Treatment with mitoxantrone, teriflunomide, fingolimod, natalizumab, azathioprine, cyclosporine, methotrexate or mycophenolate mofetil 1 year prior to baseline
* Any prior treatment with cladribine, cyclophosphamide, total lymphoid irradiation, T cell or T cell receptor products, or any therapeutic monoclonal antibody, except natalizumab
* Previous treatment with any other MS investigational drug 1 year prior to screening
* All non-MS investigational drugs must have a minimum washout of 30 days prior to screening or 5 half-lives, whatever is the longest period of time.
* HIV or hepatitis infection
* History of cancer
* Any other significant medical condition that, in the opinion of the investigator, could cause CNS tissue damage or limit its repair.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 183 (Actual)
Dates: Start 2012-08; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Brain Atrophy | 2 Years
  The percentage of brain volume change (atrophy) as measured on 24 month MRIs calculated by the central MRI facility.

SECONDARY OUTCOMES:
Disease Progression | 2 Years
  The percentage of subjects with sustained progression with definitions of sustained effect at 3 months and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Jackson, Study Director — Opexa Therapeutics, Inc.
Locations (36):
- United States (33):
  - HOPE Research Institute, Phoenix, Arizona
  - Northwest NeuroSpecialists, LLC, Tucson, Arizona
  - Alta Bates Summit Medical Center, The Research and Education Development Institute, Berkeley, California
  - Neurology Associates, P.A., Maitland, Florida
  - University of Miami, Miami, Florida
  - Collier Neurologic Specialists, LLC, Naples, Florida
  - Neurological Services of Orlando, Orlando, Florida
  - Meridien Research, Tampa, Florida
  - Vero Beach Neurology, Vero Beach, Florida
  - Shepherd Center, Atlanta, Georgia
  - Consultants In Neurology, Ltd., Northbrook, Illinois
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - Josephson Wallack Munshower Neurology, PC, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Associates in Neurology, Lexington, Kentucky
  - Saint Elizabeth's Medical Center, Boston, Massachusetts
  - Island Neurological Assoicates, PC, Plainview, New York
  - University Hospital and Medical Center Stony Brook New York, Stony Brook, New York
  - The Neurological Institute, PA, Charlotte, North Carolina
  - Carolinas Medical Center Neurology, Charlotte, North Carolina
  - PMG Research of Charlotte, Charlotte, North Carolina
  - Neurology Specialists, Inc, Dayton, Ohio
  - Providence Medical Group - Medford, Medford, Oregon
  - Providence St. Vincent Medical Center - Northwest MS Center, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - The Maxine Mesinger MS Clinic/Baylor College of Medicine, Houston, Texas
  - Central Texas Neurology, Round Rock, Texas
  - Integra Clinical Research, LLC, San Antonio, Texas
  - Fletcher Allen Health Care - Neurology Service, Burlington, Vermont
  - Hampton Roads Neurology, Newport News, Virginia
  - Neurological Associates, Inc, Richmond, Virginia
  - Swedish Neuroscience Institute, Issaquah, Washington
  - Swedish Neuroscience Institute, Seattle, Washington
- Canada (3):
  - University of Ottawa, Ottawa, Ontario
  - Recherche Sepmus Inc., Greenfield Park, Quebec
  - Montreal Neurological Institute and Hospital, Montreal, Quebec

REFERENCES:
- See also: Click here for more information about MS and current research. — http://www.nationalmssociety.org